CLINICAL TRIAL: NCT02709902
Title: A Multi-center, Double-blind, Randomized, Placebo, Controlled, Parallel-group Study, Comparing Adapalene/BP Gel, 0.3%/2.5% to EPIDUO® FORTE GEL and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: Study Comparing Adapalene/BP Gel to EPIDUO® FORTE and Both to a Placebo Control in Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADBG 1519
Record Dates: First submitted 2016-03-08; First posted 2016-03-16 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adapalene/BP gel, 0.3%/2.5% (Experimental): Topical, once daily, for 84 days.
  Interventions: Drug: Adapalene/BP gel, 0.3%/2.5%
- EPIDUO® FORTE (Active Comparator): Topical, once daily, for 84 days.
  Interventions: Drug: EPIDUO® FORTE
- Placebo (Placebo Comparator): Topical, once daily, for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adapalene/BP gel, 0.3%/2.5% — Gel
  Other Names: Adapalene, benzoyl peroxide
  Arms: Adapalene/BP gel, 0.3%/2.5%
Drug: EPIDUO® FORTE — Gel
  Other Names: Adapalene, benzoyl peroxide
  Arms: EPIDUO® FORTE
Drug: Placebo — Gel
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
Bioequivalence with Clinical Endpoints.

DETAILED DESCRIPTION:
Randomized, Double-Blind, Placebo-Controlled, Multiple-Site, Parallel Design, Bioequivalence with Clinical Endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 12 and ≤ 40years with a clinical diagnosis of acne vulgaris.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 460 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | Week 12
  Percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts
Change in non-inflammatory lesion counts | Week 12
  Percent change from baseline to week 12 in the non-inflammatory (open and closed comedones) lesion counts

SECONDARY OUTCOMES:
Clinical response of success | Week 12
  The proportion of subjects with a clinical response of success at week 12, success defined as an Investigator's Global Assessment score that is at least two grades less than the baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No